CLINICAL TRIAL: NCT07162844
Title: Effectiveness of Liquid Versus Foam Sclerotherapy With or Without Herbal Gel in Treating Telangiectasia and Reticular Veins: A Randomized Controlled Trial
Brief Title: Foam and Liquid Sclerotherapy With or Without Herbal Gel for Small Vein Treatment
Acronym: ELF-HTR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Gaheed, director, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-348; KFSIRB200-348 (Other: the scientific research committee of kafrelsheikh university)
Record Dates: First submitted 2025-08-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Telangectasia; Reticular Veins
Keywords: Telangectasia; Reticular veins; foam; Sclerotherapy; C1; liquid; varicose

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel-group clinical trial with four intervention arms. Eligible participants will be randomly assigned to receive one of the following treatments: foam polidocanol alone, liquid polidocanol alone, foam polidocanol combined with herbal gel, or liquid polidocanol combined with herbal gel. Each participant will receive only the assigned intervention throughout the study. The parallel assignment model allows for independent comparison of treatment efficacy and safety between the four groups.
Masking Description: Due to the visible and physical differences between foam and liquid polidocanol, as well as the use of adjunctive herbal gel in some arms, masking of participants and investigators was not feasible. Therefore, the study is conducted as an open-label trial with no blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- liquid sclerotherapy injection without application of herbal gel after procedure (Experimental): Participants in this group will receive liquid polidocanol injection sclerotherapy without herbal gel application
  Interventions: Procedure: Liquid sclerotherapy in telangectasia and reticular veins without application of herbal gel post procedure
- liquid sclerotherapy injection with application of herbal gel after procedure (Experimental): Participants in this group will receive liquid polidocanol injection sclerotherapy, followed by the application of a herbal gel topically at the injection site. The gel is applied immediately post-procedure twice daily
  Interventions: Procedure: Liquid sclerotherapy in telangectasia and reticular veins wit application of herbal gel post procedure
- foam sclerotherapy injection without application of herbal gel after procedure (Experimental): Participants in this group will receive foam polidocanol injection sclerotherapy without application of herbal gel
  Interventions: Procedure: foam sclerotherapy in telangectasia and reticular veins without application of herbal gel post procedure
- foam sclerotherapy injection with application of herbal gel after procedure (Experimental): Participants in this group will receive foam polidocanol injection sclerotherapy, followed by the application of a herbal gel topically at the injection site. The gel is applied immediately post-procedure twice daily
  Interventions: Procedure: foam sclerotherapy in telangectasia and reticular veins with application of herbal gel post procedure

INTERVENTIONS:
Procedure: Liquid sclerotherapy in telangectasia and reticular veins without application of herbal gel post procedure — Liquid sclerotherapy injection of polidocanol in telangectasia and reticular veins without application of herbal gel post procedure
  Arms: liquid sclerotherapy injection without application of herbal gel after procedure
Procedure: Liquid sclerotherapy in telangectasia and reticular veins wit application of herbal gel post procedure — Liquid sclerotherapy injection of polidocanol in telangectasia and reticular veins with application of herbal gel post procedure
  Arms: liquid sclerotherapy injection with application of herbal gel after procedure
Procedure: foam sclerotherapy in telangectasia and reticular veins without application of herbal gel post procedure — foam sclerotherapy injection of polidocanol in telangectasia and reticular veins without application of herbal gel post procedure
  Arms: foam sclerotherapy injection without application of herbal gel after procedure
Procedure: foam sclerotherapy in telangectasia and reticular veins with application of herbal gel post procedure — foam sclerotherapy injection of polidocanol in telangectasia and reticular veins with application of herbal gel post procedure
  Arms: foam sclerotherapy injection with application of herbal gel after procedure

SUMMARY:
Telangiectasias (spider veins) and reticular veins represent early and common manifestations of chronic venous insufficiency . Telangiectasias are dilated intradermal venules or capillaries less than 1 mm in diameter and typically appear on the thighs, calves, or ankles in a red, pink, or purple hue. Reticular veins, measuring 1-3 mm, are dilated subdermal veins located slightly deeper and often function as feeder veins to telangiectasias. They are commonly blue or green and may cause discomfort or cosmetic concerns.

According to the CEAP classification (Clinical-Etiology-Anatomy-Pathophysiology), telangiectasias and reticular veins fall under class C1. Chronic venous insufficiency of the lower extremities is increasingly prevalent, affecting nearly one-third of women and one-fifth of men, and can lead to symptoms such as leg fatigue, cramps, swelling, skin changes, or in advanced cases, deep vein thrombosis or pulmonary embolism. Telangiectasias are often the first visible signs of CVI and are frequently treated for cosmetic purposes.

Sclerotherapy is a well-established treatment for C1 venous disease. It involves the injection of a sclerosant agent into abnormal veins, causing endothelial damage, inflammation, and eventual fibrosis and closure of the vein. Among the most commonly used sclerosants are detergent-type agents like sodium tetradecyl sulfate (STS) and polidocanol (POL), which have been used effectively in both liquid and foam forms.

Liquid sclerotherapy has been employed for over 160 years, offering a minimally invasive approach to treat superficial veins. Foam sclerotherapy, introduced by Orbach and further popularized in recent decades, involves mixing the sclerosant with air or gas to form a microbubble foam. This form has increased surface area contact with the endothelium, potentially enhancing efficacy, particularly in larger veins. However, debate remains regarding the relative safety and effectiveness of foam versus liquid sclerotherapy, especially for small vessels such as telangiectasias and reticular veins.

Several clinical studies, including those by Kaygin and Halici, have compared foam and liquid sclerotherapy in treating lower limb varicose veins. Both forms have demonstrated efficacy and acceptable safety profiles. Nonetheless, further research is needed to determine the optimal form of sclerotherapy, especially in relation to cosmetic outcomes, pain, patient satisfaction, and side effect profiles. This study aims to compare the effectiveness and safety of liquid versus foam sclerotherapy, with or without herbal application in the treatment of telangiectasias and reticular veins.

DETAILED DESCRIPTION:
Telangiectasias, also known as spider veins, are dilated intradermal venules less than 1 mm in diameter. They often appear close to the surface of the skin in a tree-like pattern and may be red, blue, or purple. Spider veins are commonly located on the thighs, calves, or ankles and are primarily of cosmetic concern.

Reticular veins are slightly larger, measuring 1-3 mm in diameter, and are located just beneath the skin surface. They are bluish or greenish in color and often act as feeder veins to telangiectasias. Reticular veins are commonly found on the legs but can also appear on the face, breasts, or knees. While they do not typically protrude like varicose veins, they may cause discomfort or pain and contribute to an unattractive marbled skin appearance.

Both telangiectasias and reticular veins are classified as C1 disease within the CEAP (Clinical, Etiological, Anatomical, Pathophysiological) classification of chronic venous disorders. Chronic venous insufficiency is associated with dilatation of lower extremity veins, impaired venous return, and abnormal blood stasis. It is a common condition affecting a significant proportion of both men and women, and may be associated with symptoms such as swelling, fatigue, cramps, and restless legs. If left untreated, it can progress to more serious complications, including venous thrombosis.

Sclerotherapy is a well-established treatment for telangiectasias and reticular veins. It involves injection of a sclerosant solution into the affected veins, leading to endothelial damage, inflammation, and fibrosis. Historically, liquid sclerotherapy has been in use for over 160 years. More recently, foam sclerotherapy was developed to enhance the contact between sclerosant and the vein wall, potentially improving efficacy. Both liquid and foam sclerotherapy are considered safe and effective, though their comparative advantages remain under investigation.

Herbal gels with anti-inflammatory and venotonic properties have been explored as adjuvant therapies in the treatment of superficial venous disease. These may help reduce post-procedural symptoms, improve patient comfort, and enhance cosmetic results. However, clinical evidence regarding their effectiveness in combination with liquid or foam sclerotherapy is limited.

Rationale Telangiectasias and reticular veins represent a prevalent form of chronic venous disease with both cosmetic and symptomatic impact. While sclerotherapy is the primary treatment, the relative benefits of foam versus liquid sclerotherapy, as well as the potential added value of herbal gels, remain uncertain. A randomized controlled trial is therefore warranted to compare these approaches and evaluate their clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* telangiectasis on thigh or leg side
* Competent saphenofemoral and saphenopoliteal junction
* Patient post surgical stripping or post thermal ablation
* clinical classification of chronic venous disease C1(mild venous disease), -
* minimum age of 18 year-old and maximum age 65 year-old -

Exclusion Criteria:

* varicose disease in any quantity or location with clinical classification of chronic venous
* disease different of C1(mild venous disease)
* arterial insufficiency
* patient allergic to the sclerosant material or herbal gel
* dermatitis on application site
* patient with serious comorbidities like heart failure, respiratory failure, - uncontrolled hypertension with medication, and uncontrolled hypothyroidism - pregnancy - previous deep vein thrombosis (DVT) - family history of DVT - thrombophilia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Appearance of Telangiectasia and Reticular Veins Assessed by the Physician and Patient Global Assessment Scale | 4 weeks
  Improvement from baseline in appearance of telangiectasia and reticular veins, assessed using a 5-point Global Assessment Scale (0 = no improvement, 4 = complete resolution). Both physician and patient will provide independent scores.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | 4 weeks after treatment
  Incidence of adverse events including hyperpigmentation, bruising, allergic reaction, and anaphylaxis, assessed through clinical examination and patient report.

CONTACTS AND LOCATIONS:
Overall Officials: moustafa hassan mabrouk, lecturer, Study Director — faculty of medicine kfs university
Locations (1):
- Faculty of medicine kfs university, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes